CLINICAL TRIAL: NCT01945021
Title: Phase II, Open Label, Single Arm Study of the Efficacy and Safety of Crizotinib in East Asian Patients With Advanced ALK-Negative NSCLC Harboring a Translocation or Inversion Involving the c-ROS Oncogene (ROS1) Locus
Brief Title: Phase II Safety and Efficacy Study of Crizotinib in East Asian Patients With ROS1 Positive, ALK Negative Advanced NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: OxOnc Development LP (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OO 12-01
Record Dates: First submitted 2013-09-05; First posted 2013-09-18 (Estimated); Results first posted 2016-08-01 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Non Small Cell Lung Cancer; ROS1 Proto Oncogene; Crizotinib
Keywords: Non small cell lung cancer; NSCLC; ROS1; ROS1 positive; ROS1 proto oncogene; c ros tyrosine kinases; ROS1 positive NSCLC; ROS1 lung cancer; ALK negative; Lung Carcinoma; Neoplasm; Crizotinib; Xalkori; Previously treated or untreated; North East Asian
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Neoplasms | interventions — Crizotinib

ARMS (1):
- Crizotinib (Experimental): Single-arm trial whereby all consented, enrolled, eligible patients receive crizotinib
  Interventions: Drug: Crizotinib

INTERVENTIONS:
Drug: Crizotinib
  Other Names: Xalkori

SUMMARY:
To assess treatment effectiveness and safety of oral crizotinib administered to East Asian patients with Advanced Non-Small Cell Lung Cancer (NSCLC) that is confirmed to be positive for a ROS1 positive gene mutation (translocation or inversion) and confirmed negative for an ALK mutation

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis of NSCLC that is locally advanced or metastatic
* treatment-naïve or have received no more than 3 systemic treatment regimen(s)
* Positive for translocation or inversion events involving the ROS1 gene
* Negative for translocation or inversion events involving the ALK gene
* Patients with brain metastases are eligible if asymptomatic, or if treated, must be neurologically stable for at least 2 weeks and are not taking any contraindicated medications
* Any prior treatment (chemotherapy, radiation [except for palliative], or surgery) must have been completed at least 2 weeks prior to initiation of study medication
* At least 1 measurable tumor lesion as per RECIST v1.1
* Female or male, 18 years of age or older
* ECOG performance status 0 to 1
* Adequate organ function
* Signed and dated informed consent
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures, including completion of the PRO measures
* Agree to use effective contraception during the study period and for at least 90 days after completion of the study treatment

Exclusion Criteria:

* Current treatment on another therapeutic clinical trial
* Prior therapy specifically directed against ALK or ROS1 fusion genes
* Spinal cord compression unless treated with the patient attaining good pain control and stable or recovered neurologic function, carcinomatous meningitis, or leptomeningeal disease
* known interstitial fibrosis or interstitial lung disease
* myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, or cerebrovascular accident including transient ischemic attack within 3 months prior to start of study treatment
* Ongoing cardiac dysrhythmias of NCI CTCAE v4.03 Grade >/=2, uncontrolled atrial fibrillation of any grade, or QTc >470 msec
* Pregnant or breast feeding
* Use of drugs or foods that are known potent CYP3A4 inhibitors or inducers
* Use of other anti-cancer drugs including traditional Chinese medicine on the SFDA list
* Evidence of active malignancy within last 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2013-09-30 (Actual); Primary Completion 2015-07-31 (Actual); Study Completion 2020-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (44):
- China (25):
  - The First Affiliated Hospital of Anhui Medical University, Department of Medical Oncology, Hefei, Anhui
  - Department of Medical Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Chaoyang District, Beijing Municipality
  - The Military General Hospital of Beijing PLA / Medical Oncology Dept., Dongcheng District, Beijing Municipality
  - 307 Hospital of PLA/Department of Lung Cancer, Fengtai District, Beijing Municipality
  - Beijing Cancer Hospital, Department of Thoracic Oncology, Haidian District, Beijing Municipality
  - Chinese PLA General Hospital, Haidian District, Beijing Municipality
  - Beijing Chest Hospital, Tongzhou District, Beijing Municipality
  - Respiration department,the First Affiliated Hospital of Third Military Medical University, PLA, Shapingba District, Chongqing Municipality
  - Fujian Province Oncology Hospital, Fuzhou, Fujian
  - SUN Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Hunan Provincial Tumor Hospital/Division of Oncology, Changsha, Hunan
  - Department of Oncology, Jilin Provincial Cancer Hospital, Changchun, Jilin
  - The affiliated hospital of medical college Qingdao University / Medical oncology department, Qingdao, Shandong
  - Department of Pulmonary Medicine, Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital/Lung cancer clinical center, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University / Respiratory Department, Xuhui District, Shanghai Municipality
  - Oncology Department, West China Hospital of Sichuan University, Chengdu, Sichuan
  - Sichuan Province Cancer Hospital/Department of Pulmonary Tumor, Chengdu, Sichuan
  - Department of Thoracic Oncology, Tianjin Medical University Cancer Institute and Hospital, Hexi District, Tianjin Municipality
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital of College of Medicine of Zhejiang University, Center for Oncology, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
- Japan (11):
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - Aichi Cancer Center Hospital, Aichi
  - National Cancer Center Hospital East, Chiba
  - NHO Shikoku Cancer Center, Ehime
  - NHO Kyushu Cancer Center, Fukuoka
  - Hyogo Cancer Center, Hyōgo
  - Tohoku University Hospital, Miyagi
  - Kinki University Hospital, Osaka
  - Osaka City General Hospital, Osaka
  - Cancer Institute Hospital of JFCR, Tokyo
  - National Cancer Center Hospital, Tokyo
- South Korea (4):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Yonsei University, Severance Hospital, Seoul
- Taiwan (4):
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

REFERENCES:
- [Derived] Wu YL, Yang JC, Kim DW, Lu S, Zhou J, Seto T, Yang JJ, Yamamoto N, Ahn MJ, Takahashi T, Yamanaka T, Kemner A, Roychowdhury D, Paolini J, Usari T, Wilner KD, Goto K. Phase II Study of Crizotinib in East Asian Patients With ROS1-Positive Advanced Non-Small-Cell Lung Cancer. J Clin Oncol. 2018 May 10;36(14):1405-1411. doi: 10.1200/JCO.2017.75.5587. Epub 2018 Mar 29. PMID 29596029

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 129 participants with anaplastic lymphoma kinase (ALK) negative advanced non-small cell lung cancer (NSCLC) harboring a translocation or inversion event involving the c-ros oncogene 1 (ROS1) locus were enrolled of whom 127 were allocated to treatment with crizotinib and 2 participants had screen failures.
Groups:
- Crizotinib 250 mg: Participants received crizotinib 250 mg orally twice a day in a cycle of 28 days. Dose was modified by investigator if there was treatment-related toxicity. Maximum treatment exposure time was of 291.9 weeks up to final analysis date.
Period: Overall Study
Arm/Group | Crizotinib 250 mg
Started | 127
Safety Population | 127 (Received at least 1 dose of study medication.)
Response Evaluable Population | 127 (Received at least 1 dose of study drug and an adequate baseline tumor assessment.)
Patient Reported Outcome Evaluable | 123 (Received at least 1 dose of study drug, completed baseline with at least 1 post-baseline assessment.)
Completed | 44
Not Completed | 83
Not completed — Adverse Event | 1
Not completed — Withdrawal of consent | 12
Not completed — Lost to Follow-up | 5
Not completed — Death | 65

BASELINE CHARACTERISTICS:
Population: The Safety Population contains all enrolled participants who received at least one dose of study medication.
Arm/Group | Crizotinib 250 mg
Number analyzed (Participants) | 127
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.48 (12.136)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73
  Male | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 127
Region of Enrollment [Count of Participants; unit: Participants]
  Asia: China | 74
  Asia: Japan | 26
  Asia: Korea | 12
  Asia: Taiwan | 15

OUTCOME MEASURES:

1. Primary Outcome: Independent Radiology Reviewed Overall Objective Response (ORR)
Description: Overall objective response (ORR) was defined as the number of patients with a best overall response of confirmed Complete Response or confirmed Partial Response according to RECIST v1.1 (as determined by Independent Radiology Review [IRR]), relative to the total population of response-evaluable participants. Per RECIST v1.1, CR: disappearance of all target lesions. Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis); PR: at least 30% decrease in sum of diameters of target lesions, taking as reference baseline sum diameters. Confirmed responses were those that persisted on repeat imaging at least 4 weeks after the initial documentation of response.
Time Frame: Starting from the first dose study treatment until the first documented CR or PR (every 8 weeks then after 8 cycles at every 12 weeks in duration of 94.0 weeks)
Population: The response-evaluable population (RES) population included all enrolled participants who received at least 1 dose of study medication and had an adequate baseline tumor assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib 250 mg
Number analyzed (Participants) | 127
Participants | 88

2. Secondary Outcome: IRR-Assessed Duration of Response (DR)
Description: DR: time from first documentation of objective tumor response (CR or PR) to first documentation of objective progressive disease (PD) or to death due to any cause, whichever occurred first. If no progression or death on study was observed, or given antitumor treatment other than study drug, participants were censored on date of last on-study tumor assessment. RECIST v1.1, a) PD: >=20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study (this includes baseline sum if that is the smallest on study), sum must also demonstrate an absolute increase of >=5 mm, appearance of 1 or more new lesions, unequivocal progression of existing non-target lesions; b) CR: disappearance of all target lesions. Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis); c) PR: >=30% decrease in sum of diameters of target lesions, taking as reference baseline sum diameters.
Time Frame: From first documentation of objective tumor response to first documentation of objective PD or death due to any cause, whichever occurred first (every 8 weeks then after 8 cycles at every 12 weeks in duration of 151.3 weeks)
Population: The RES population included all enrolled participants who received at least 1 dose of study medication and had an adequate baseline tumor assessment. Here, "Overall Number of Participants Analyzed" signifies number of participants with a confirmed objective response that could have occurred anytime up to 151.3 weeks.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Crizotinib 250 mg
Number analyzed (Participants) | 91
Months | 19.7 [14.1 to NA] — Upper limit cannot be estimated due to less number of participants with event.

3. Secondary Outcome: IRR-Assessed Time to Tumor Response (TTR)
Description: TTR was defined as the time from the date of first dose to first documentation of objective tumor response (CR or PR), that was subsequently confirmed. For participants proceeding from PR to CR, the onset of PR was taken as the onset of response. RECIST v1.1 (as determined by IRR), a) CR: disappearance of all target lesions. Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis); b) PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From date of first dose of crizotinib to first documentation of objective response was observed (every 8 weeks then after 8 cycles at every 12 weeks in duration of 151.3 weeks)
Population: as for outcome 2
Measure: Median (Full Range); unit: Months
Arm/Group | Crizotinib 250 mg
Number analyzed (Participants) | 91
Months | 1.9 [1.6 to 15.8]

4. Secondary Outcome: IRR Assessed Disease Control Rate (DCR) at 8 Weeks
Description: DCR at 8 weeks was defined as the percentage of participants with a confirmed CR, confirmed PR, or stable disease (SD) at 8 weeks, respectively, relative to the total population of response evaluable participants. RECIST v1.1 (as determined by IRR), a) CR: disappearance of all target lesions. Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis); b) PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: At 8 weeks after the start of study treatment
Population: The RES population included all enrolled participants who received at least 1 dose of study medication and had an adequate baseline tumor assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Crizotinib 250 mg
Number analyzed (Participants) | 127
Percentage of participants | 88.2 [81.3 to 93.2]

5. Secondary Outcome: IRR-Assessed Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of the first dose of crizotinib to first documentation of objective PD or to death on study due to any cause, whichever occurred first. If no progression or death on study was observed, or given antitumor treatment other than study drug, participants were censored on date of last on-study tumor assessment. RECIST v1.1, PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered a sign of progression. Unequivocal progression of existing non-target lesions.
Time Frame: From the date of first dose of crizotinib until the first documentation of objective PD or death (every 8 weeks then after 8 cycles at every 12 weeks in duration of 151.3 weeks)
Population: The safety analysis population (SAF) included all enrolled participants who received at least 1 dose of study medication.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Crizotinib 250 mg
Number analyzed (Participants) | 127
Months | 15.9 [12.9 to 24.0]

6. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of the first dose of crizotinib to the date of death due to any cause. For participants still alive at the time of analysis, the OS time was censored on the last date the participants were known to be alive.
Time Frame: From date of the first dose of crizotinib until the date of death from any cause (up to 291.9 weeks)
Population: SAF included all enrolled participants who received at least 1 dose of study medication.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Crizotinib 250 mg
Number analyzed (Participants) | 127
Months | 44.2 [32.0 to NA] — Upper limit was not estimable due to high number of participants were censored.

7. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious AEs, Treatment Emergent Treatment Related AEs and SAEs, Grade 3 or 4 Treatment Emergent AEs and Grade 3 or 4 Treatment Emergent Treatment Related AEs
Description: Treatment-emergent AEs :between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to crizotinib was assessed by the investigator. Treatment-related AE: any untoward medical occurrence attributed to study drug in a participant who received study drug. Serious adverse event (SAE):an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Grade 3 (Severe) events=unacceptable or intolerable events, significantly interrupting usual daily activity, require systemic drug therapy/other treatment. Grade 4 (Life-threatening) events caused participant to be in imminent danger of death.
Time Frame: Baseline up to 28 days after the last dose of study treatment (maximum up to 295.9 weeks)
Population: SAF included all enrolled participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib 250 mg
Number analyzed (Participants) | 127
Participants
  Incidence of All-Causality Adverse Events | 127
  Incidence of All-Causality Serious Adverse Events | 46
  Incidence of Treatment Related Adverse Events | 124
  Incidence of Treatment Related Serious Adverse Events | 11
  Incidence of All-Causality Grade 3-4 Adverse Event | 68
  Incidence of Treatment Related Grade 3-4 Adverse Event | 41

8. Secondary Outcome: Number of Participants With a Shift in Hematology Laboratory Results From Baseline Grade </=2 to Worst Grade 3 or Grade 4
Description: Laboratory values included hemoglobin increased, anemia, platelet count decreased, leukocytosis, white blood cell decreased, lymphocyte count increased, lymphocyte count decreased and neutrophil count decreased. Laboratory values were defined as National Cancer Institute Common Toxicity Criteria for Adverse Events Version 3.0 (NCI CTCAE v3.0) grade 3 or higher.
Time Frame: Baseline up to 28 days after the last dose of study treatment (maximum up to 295.9 weeks)
Population: SAF included all enrolled participants who received at least 1 dose of study medication. Here, "number analyzed" signifies participants evaluable at specific rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib 250 mg
Number analyzed (Participants) | 127
Participants
  Hemoglobin Increased: Baseline Grade 0 to Worst Grade 3 | 0
  Hemoglobin Increased: Baseline Grade 1 to Worst Grade 3 | 0
  Hemoglobin Increased: Baseline Grade 2 to Worst Grade 3 | 0
  Hemoglobin Increased: Baseline Grade 0 to Worst Grade 4: number analyzed (Participants) | 0
  Hemoglobin Increased: Baseline Grade 1 to Worst Grade 4: number analyzed (Participants) | 0
  Hemoglobin Increased: Baseline Grade 2 to Worst Grade 4: number analyzed (Participants) | 0
  Anemia: Baseline Grade 0 to Worst Grade 3 | 2
  Anemia: Baseline Grade 1 to Worst Grade 3 | 1
  Anemia: Baseline Grade 2 to Worst Grade 3 | 5
  Anemia: Baseline Grade 0 to Worst Grade 4 | 0
  Anemia: Baseline Grade 1 to Worst Grade 4 | 0
  Anemia: Baseline Grade 2 to Worst Grade 4 | 0
  Platelet Count Decreased: Baseline Grade 0 to Worst Grade 3 | 0
  Platelet Count Decreased: Baseline Grade 1 to Worst Grade 3 | 0
  Platelet Count Decreased: Baseline Grade 2 to Worst Grade 3 | 0
  Platelet Count Decreased: Baseline Grade 0 to Worst Grade 4 | 0
  Platelet Count Decreased: Baseline Grade 1 to Worst Grade 4 | 0
  Platelet Count Decreased: Baseline Grade 2 to Worst Grade 4 | 0
  Leukocytosis: Baseline Grade 0 to Worst Grade 3 | 0
  Leukocytosis: Baseline Grade 1 to Worst Grade 3: number analyzed (Participants) | 0
  Leukocytosis: Baseline Grade 2 to Worst Grade 3: number analyzed (Participants) | 0
  Leukocytosis: Baseline Grade 0 to Worst Grade 4 | 0
  Leukocytosis: Baseline Grade 1 to Worst Grade 4: number analyzed (Participants) | 0
  Leukocytosis: Baseline Grade 2 to Worst Grade 4: number analyzed (Participants) | 0
  White Blood Cell Decreased: Baseline Grade 0 to Worst Grade 3 | 3
  White Blood Cell Decreased: Baseline Grade 1 to Worst Grade 3 | 1
  White Blood Cell Decreased: Baseline Grade 2 to Worst Grade 3 | 0
  White Blood Cell Decreased: Baseline Grade 0 to Worst Grade 4 | 0
  White Blood Cell Decreased: Baseline Grade 1 to Worst Grade 4 | 0
  White Blood Cell Decreased: Baseline Grade 2 to Worst Grade 4 | 0
  Lymphocyte Count Increased: Baseline Grade 0 to Worst Grade 3: number analyzed (Participants) | 83
  Lymphocyte Count Increased: Baseline Grade 0 to Worst Grade 3 | 0
  Lymphocyte Count Increased: Baseline Grade 1 to Worst Grade 3: number analyzed (Participants) | 0
  Lymphocyte Count Increased: Baseline Grade 2 to Worst Grade 3: number analyzed (Participants) | 83
  Lymphocyte Count Increased: Baseline Grade 2 to Worst Grade 3 | 0
  Lymphocyte Count Increased: Baseline Grade 0 to Worst Grade 4: number analyzed (Participants) | 0
  Lymphocyte Count Increased: Baseline Grade 1 to Worst Grade 4: number analyzed (Participants) | 0
  Lymphocyte Count Increased: Baseline Grade 2 to Worst Grade 4: number analyzed (Participants) | 0
  Lymphocyte Count Decreased: Baseline Grade 0 to Worst Grade 3: number analyzed (Participants) | 83
  Lymphocyte Count Decreased: Baseline Grade 0 to Worst Grade 3 | 4
  Lymphocyte Count Decreased: Baseline Grade 1 to Worst Grade 3: number analyzed (Participants) | 83
  Lymphocyte Count Decreased: Baseline Grade 1 to Worst Grade 3 | 0
  Lymphocyte Count Decreased: Baseline Grade 2 to Worst Grade 3: number analyzed (Participants) | 83
  Lymphocyte Count Decreased: Baseline Grade 2 to Worst Grade 3 | 2
  Lymphocyte Count Decreased: Baseline Grade 0 to Worst Grade 4: number analyzed (Participants) | 83
  Lymphocyte Count Decreased: Baseline Grade 0 to Worst Grade 4 | 0
  Lymphocyte Count Decreased: Baseline Grade 1 to Worst Grade 4: number analyzed (Participants) | 83
  Lymphocyte Count Decreased: Baseline Grade 1 to Worst Grade 4 | 0
  Lymphocyte Count Decreased: Baseline Grade 2 to Worst Grade 4: number analyzed (Participants) | 83
  Lymphocyte Count Decreased: Baseline Grade 2 to Worst Grade 4 | 0
  Neutrophil Count Decreased: Baseline Grade 0 to Worst Grade 3: number analyzed (Participants) | 101
  Neutrophil Count Decreased: Baseline Grade 0 to Worst Grade 3 | 7
  Neutrophil Count Decreased: Baseline Grade 1 to Worst Grade 3: number analyzed (Participants) | 101
  Neutrophil Count Decreased: Baseline Grade 1 to Worst Grade 3 | 1
  Neutrophil Count Decreased: Baseline Grade 2 to Worst Grade 3: number analyzed (Participants) | 101
  Neutrophil Count Decreased: Baseline Grade 2 to Worst Grade 3 | 0
  Neutrophil Count Decreased: Baseline Grade 0 to Worst Grade 4: number analyzed (Participants) | 101
  Neutrophil Count Decreased: Baseline Grade 0 to Worst Grade 4 | 4
  Neutrophil Count Decreased: Baseline Grade 1 to Worst Grade 4: number analyzed (Participants) | 101
  Neutrophil Count Decreased: Baseline Grade 1 to Worst Grade 4 | 0
  Neutrophil Count Decreased: Baseline Grade 2 to Worst Grade 4: number analyzed (Participants) | 101
  Neutrophil Count Decreased: Baseline Grade 2 to Worst Grade 4 | 0

9. Secondary Outcome: Number of Participants With a Shift of Chemistry Laboratory Results From Baseline Grade </=2 to Worst Grade 3 or Grade 4
Description: Laboratory values included blood bilirubin increased, alanine aminotransferase increased, aspartate aminotransferase increased, alkaline phosphatase increased, hypoalbuminemia, hypernatremia, hyponatremia, hyperkalemia, hypokalemia, hypercalcemia, hypocalcemia, hypophosphatemia, Creatinine increased, hyperuricemia, hypermagnesemia, hypomagnesemia, hyperglycemia and hypoglycemia. Laboratory values were defined as National Cancer Institute Common Toxicity Criteria for Adverse Events Version 3.0 (NCI CTCAE v3.0) grade 3 or higher.
Time Frame: Baseline up to 28 days after the last dose of study treatment (maximum up to 295.9 weeks)
Population: SAF included all enrolled participants who received at least one dose of study medication. Here, "number analyzed" signifies participants evaluable at specific rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib 250 mg
Number analyzed (Participants) | 127
Participants
  Blood Bilirubin Increased: Baseline Grade 0 to Worst Grade 3 | 1
  Blood Bilirubin Increased: Baseline Grade 1 to Worst Grade 3 | 0
  Blood Bilirubin Increased: Baseline Grade 2 to Worst Grade 3 | 0
  Blood Bilirubin Increased: Baseline Grade 0 to Worst Grade 4 | 0
  Blood Bilirubin Increased: Baseline Grade 1 to Worst Grade 4 | 0
  Blood Bilirubin Increased: Baseline Grade 2 to Worst Grade 4 | 0
  Alanine Aminotransferase Increased: Baseline Grade 0 to Worst Grade 3 | 4
  Alanine Aminotransferase Increased: Baseline Grade 1 to Worst Grade 3 | 1
  Alanine Aminotransferase Increased: Baseline Grade 2 to Worst Grade 3 | 0
  Alanine Aminotransferase Increased: Baseline Grade 0 to Worst Grade 4 | 4
  Alanine Aminotransferase Increased: Baseline Grade 1 to Worst Grade 4 | 0
  Alanine Aminotransferase Increased: Baseline Grade 2 to Worst Grade 4 | 0
  Aspartate Aminotransferase Increased : Baseline Grade 0 to Worst Grade 3 | 2
  Aspartate Aminotransferase Increased : Baseline Grade 1 to Worst Grade 3 | 0
  Aspartate Aminotransferase Increased : Baseline Grade 2 to Worst Grade 3 | 0
  Aspartate Aminotransferase Increased : Baseline Grade 0 to Worst Grade 4 | 4
  Aspartate Aminotransferase Increased : Baseline Grade 1 to Worst Grade 4 | 0
  Aspartate Aminotransferase Increased : Baseline Grade 2 to Worst Grade 4 | 0
  Alkaline Phosphatase Increased : Baseline Grade 0 to Worst Grade 3 | 0
  Alkaline Phosphatase Increased : Baseline Grade 1 to Worst Grade 3 | 0
  Alkaline Phosphatase Increased : Baseline Grade 2 to Worst Grade 3 | 0
  Alkaline Phosphatase Increased : Baseline Grade 0 to Worst Grade 4 | 0
  Alkaline Phosphatase Increased : Baseline Grade 1 to Worst Grade 4 | 0
  Alkaline Phosphatase Increased : Baseline Grade 2 to Worst Grade 4 | 0
  Hypoalbuminemia: Baseline Grade 0 to Worst Grade 3 | 1
  Hypoalbuminemia: Baseline Grade 1 to Worst Grade 3 | 1
  Hypoalbuminemia: Baseline Grade 2 to Worst Grade 3 | 1
  Hypoalbuminemia: Baseline Grade 0 to Worst Grade 4 | 0
  Hypoalbuminemia: Baseline Grade 1 to Worst Grade 4 | 0
  Hypoalbuminemia: Baseline Grade 2 to Worst Grade 4 | 0
  Hypernatremia: Baseline Grade 0 to Worst Grade 3 | 0
  Hypernatremia: Baseline Grade 1 to Worst Grade 3 | 0
  Hypernatremia: Baseline Grade 2 to Worst Grade 3 | 0
  Hypernatremia: Baseline Grade 0 to Worst Grade 4 | 0
  Hypernatremia: Baseline Grade 1 to Worst Grade 4 | 0
  Hypernatremia: Baseline Grade 2 to Worst Grade 4 | 0
  Hyponatremia: Baseline Grade 0 to Worst Grade 3 | 8
  Hyponatremia: Baseline Grade 1 to Worst Grade 3 | 4
  Hyponatremia: Baseline Grade 2 to Worst Grade 3: number analyzed (Participants) | 0
  Hyponatremia: Baseline Grade 0 to Worst Grade 4 | 0
  Hyponatremia: Baseline Grade 1 to Worst Grade 4 | 0
  Hyponatremia: Baseline Grade 2 to Worst Grade 4: number analyzed (Participants) | 0
  Hyperkalemia: Baseline Grade 0 to Worst Grade 3 | 0
  Hyperkalemia: Baseline Grade 1 to Worst Grade 3 | 1
  Hyperkalemia: Baseline Grade 2 to Worst Grade 3 | 0
  Hyperkalemia: Baseline Grade 0 to Worst Grade 4 | 0
  Hyperkalemia: Baseline Grade 1 to Worst Grade 4 | 0
  Hyperkalemia: Baseline Grade 2 to Worst Grade 4 | 0
  Hypokalemia: Baseline Grade 0 to Worst Grade 3 | 5
  Hypokalemia: Baseline Grade 1 to Worst Grade 3 | 0
  Hypokalemia: Baseline Grade 2 to Worst Grade 3 | 0
  Hypokalemia: Baseline Grade 0 to Worst Grade 4 | 1
  Hypokalemia: Baseline Grade 1 to Worst Grade 4 | 0
  Hypokalemia: Baseline Grade 2 to Worst Grade 4 | 0
  Hypercalcemia: Baseline Grade 0 to Worst Grade 3 | 0
  Hypercalcemia: Baseline Grade 1 to Worst Grade 3 | 0
  Hypercalcemia: Baseline Grade 2 to Worst Grade 3 | 0
  Hypercalcemia: Baseline Grade 0 to Worst Grade 4 | 0
  Hypercalcemia: Baseline Grade 1 to Worst Grade 4 | 0
  Hypercalcemia: Baseline Grade 2 to Worst Grade 4 | 0
  Hypocalcemia: Baseline Grade 0 to Worst Grade 3 | 0
  Hypocalcemia: Baseline Grade 1 to Worst Grade 3 | 0
  Hypocalcemia: Baseline Grade 2 to Worst Grade 3 | 0
  Hypocalcemia: Baseline Grade 0 to Worst Grade 4 | 0
  Hypocalcemia: Baseline Grade 1 to Worst Grade 4 | 0
  Hypocalcemia: Baseline Grade 2 to Worst Grade 4 | 0
  Hypophosphatemia: Baseline Grade 0 to Worst Grade 3: number analyzed (Participants) | 126
  Hypophosphatemia: Baseline Grade 0 to Worst Grade 3 | 11
  Hypophosphatemia: Baseline Grade 1 to Worst Grade 3: number analyzed (Participants) | 126
  Hypophosphatemia: Baseline Grade 1 to Worst Grade 3 | 0
  Hypophosphatemia: Baseline Grade 2 to Worst Grade 3: number analyzed (Participants) | 126
  Hypophosphatemia: Baseline Grade 2 to Worst Grade 3 | 1
  Hypophosphatemia: Baseline Grade 0 to Worst Grade 4: number analyzed (Participants) | 126
  Hypophosphatemia: Baseline Grade 0 to Worst Grade 4 | 1
  Hypophosphatemia: Baseline Grade 1 to Worst Grade 4: number analyzed (Participants) | 126
  Hypophosphatemia: Baseline Grade 1 to Worst Grade 4 | 0
  Hypophosphatemia: Baseline Grade 2 to Worst Grade 4: number analyzed (Participants) | 126
  Hypophosphatemia: Baseline Grade 2 to Worst Grade 4 | 0
  Creatinine Increased: Baseline Grade 0 to Worst Grade 3 | 1
  Creatinine Increased: Baseline Grade 1 to Worst Grade 3 | 0
  Creatinine Increased: Baseline Grade 2 to Worst Grade 3 | 0
  Creatinine Increased: Baseline Grade 0 to Worst Grade 4 | 0
  Creatinine Increased: Baseline Grade 1 to Worst Grade 4 | 0
  Creatinine Increased: Baseline Grade 2 to Worst Grade 4 | 0
  Hyperuricemia: Baseline Grade 0 to Worst Grade 3: number analyzed (Participants) | 126
  Hyperuricemia: Baseline Grade 0 to Worst Grade 3 | 33
  Hyperuricemia: Baseline Grade 1 to Worst Grade 3: number analyzed (Participants) | 126
  Hyperuricemia: Baseline Grade 1 to Worst Grade 3 | 0
  Hyperuricemia: Baseline Grade 2 to Worst Grade 3: number analyzed (Participants) | 0
  Hyperuricemia: Baseline Grade 0 to Worst Grade 4: number analyzed (Participants) | 126
  Hyperuricemia: Baseline Grade 0 to Worst Grade 4 | 0
  Hyperuricemia: Baseline Grade 1 to Worst Grade 4: number analyzed (Participants) | 126
  Hyperuricemia: Baseline Grade 1 to Worst Grade 4 | 0
  Hyperuricemia: Baseline Grade 2 to Worst Grade 4: number analyzed (Participants) | 0
  Hypermagnesemia: Baseline Grade 0 to Worst Grade 3: number analyzed (Participants) | 126
  Hypermagnesemia: Baseline Grade 0 to Worst Grade 3 | 2
  Hypermagnesemia: Baseline Grade 1 to Worst Grade 3: number analyzed (Participants) | 126
  Hypermagnesemia: Baseline Grade 1 to Worst Grade 3 | 0
  Hypermagnesemia: Baseline Grade 2 to Worst Grade 3: number analyzed (Participants) | 0
  Hypermagnesemia: Baseline Grade 0 to Worst Grade 4: number analyzed (Participants) | 126
  Hypermagnesemia: Baseline Grade 0 to Worst Grade 4 | 0
  Hypermagnesemia: Baseline Grade 1 to Worst Grade 4: number analyzed (Participants) | 126
  Hypermagnesemia: Baseline Grade 1 to Worst Grade 4 | 0
  Hypermagnesemia: Baseline Grade 2 to Worst Grade 4: number analyzed (Participants) | 0
  Hypomagnesemia: Baseline Grade 0 to Worst Grade 3: number analyzed (Participants) | 126
  Hypomagnesemia: Baseline Grade 0 to Worst Grade 3 | 0
  Hypomagnesemia: Baseline Grade 1 to Worst Grade 3: number analyzed (Participants) | 126
  Hypomagnesemia: Baseline Grade 1 to Worst Grade 3 | 0
  Hypomagnesemia: Baseline Grade 2 to Worst Grade 3: number analyzed (Participants) | 126
  Hypomagnesemia: Baseline Grade 2 to Worst Grade 3 | 0
  Hypomagnesemia: Baseline Grade 0 to Worst Grade 4: number analyzed (Participants) | 126
  Hypomagnesemia: Baseline Grade 0 to Worst Grade 4 | 0
  Hypomagnesemia: Baseline Grade 1 to Worst Grade 4: number analyzed (Participants) | 126
  Hypomagnesemia: Baseline Grade 1 to Worst Grade 4 | 0
  Hypomagnesemia: Baseline Grade 2 to Worst Grade 4: number analyzed (Participants) | 126
  Hypomagnesemia: Baseline Grade 2 to Worst Grade 4 | 0
  Hyperglycemia: Baseline Grade 0 to Worst Grade 3: number analyzed (Participants) | 126
  Hyperglycemia: Baseline Grade 0 to Worst Grade 3 | 1
  Hyperglycemia: Baseline Grade 1 to Worst Grade 3: number analyzed (Participants) | 126
  Hyperglycemia: Baseline Grade 1 to Worst Grade 3 | 1
  Hyperglycemia: Baseline Grade 2 to Worst Grade 3: number analyzed (Participants) | 126
  Hyperglycemia: Baseline Grade 2 to Worst Grade 3 | 0
  Hyperglycemia: Baseline Grade 0 to Worst Grade 4: number analyzed (Participants) | 126
  Hyperglycemia: Baseline Grade 0 to Worst Grade 4 | 0
  Hyperglycemia: Baseline Grade 1 to Worst Grade 4: number analyzed (Participants) | 126
  Hyperglycemia: Baseline Grade 1 to Worst Grade 4 | 0
  Hyperglycemia: Baseline Grade 2 to Worst Grade 4: number analyzed (Participants) | 126
  Hyperglycemia: Baseline Grade 2 to Worst Grade 4 | 0
  Hypoglycemia: Baseline Grade 0 to Worst Grade 3: number analyzed (Participants) | 126
  Hypoglycemia: Baseline Grade 0 to Worst Grade 3 | 0
  Hypoglycemia: Baseline Grade 1 to Worst Grade 3: number analyzed (Participants) | 126
  Hypoglycemia: Baseline Grade 1 to Worst Grade 3 | 0
  Hypoglycemia: Baseline Grade 2 to Worst Grade 3: number analyzed (Participants) | 126
  Hypoglycemia: Baseline Grade 2 to Worst Grade 3 | 0
  Hypoglycemia: Baseline Grade 0 to Worst Grade 4: number analyzed (Participants) | 126
  Hypoglycemia: Baseline Grade 0 to Worst Grade 4 | 0
  Hypoglycemia: Baseline Grade 1 to Worst Grade 4: number analyzed (Participants) | 126
  Hypoglycemia: Baseline Grade 1 to Worst Grade 4 | 0
  Hypoglycemia: Baseline Grade 2 to Worst Grade 4: number analyzed (Participants) | 126
  Hypoglycemia: Baseline Grade 2 to Worst Grade 4 | 0

10. Secondary Outcome: Change From Baseline to Cycle 60 in the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life (QOL) Questionnaire Core 30 (QLQ-C30) Scores
Description: The EORTC QLQ-C30 consists of 30 questions which are incorporated into 5 functional domains (physical, role, cognitive, emotional, and social); a global health status/global QOL scale; 3 symptom scales (fatigue, pain, nausea and vomiting scales); and 6 single items that assess the additional symptoms (dyspnea, appetite loss, sleep disturbance/insomnia, constipation, and diarrhea) and the perceived financial burden of treatment. All the scales and single-item scores ranged from 0 to 100, higher score is indicative of a higher response level (high score for a functional scale represents a high / healthy level of functioning; high score for the global health status / QoL represents a high QoL; a high score for a symptom scale / item represents a high level of symptomatology / problems).
Time Frame: Baseline up to Cycle 60
Population: Patient reported outcome (PRO)-evaluable population (PRO) included enrolled participants who received at least 1 dose of study medication and completed the assessments at baseline and with at least 1 post-baseline time point. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Crizotinib 250 mg
Number analyzed (Participants) | 26
Units on a scale
  Global Health Status | 11.85 (20.844)
  Physical Functioning | 3.08 (11.964)
  Role Functioning | -0.65 (17.945)
  Emotional Functioning | 10.77 (18.146)
  Cognitive Functioning | 3.20 (14.159)
  Social Functioning | 5.13 (20.961)
  Fatigue | -12.30 (20.156)
  Nausea and Vomiting | 0.64 (14.517)
  Pain | -12.18 (16.027)
  Dyspnea | -6.41 (21.124)
  Insomnia | -11.53 (16.161)
  Appetite loss | -14.10 (23.428)
  Constipation | 10.26 (27.920)
  Diarrhoea | 1.28 (19.937)
  Financial difficulties | -21.80 (28.199)

11. Secondary Outcome: Change From Baseline to Cycle 60 in the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Lung Cancer Module 13 Scores
Description: The EORTC QLQ-LC13 consisted of 1 multi-item scale and 9 single items that assessed specific symptoms (dyspnea, cough, hemoptysis, and site-specific pain), side effects (sore mouth, dysphagia, neuropathy, and alopecia). Scores on each scale and item ranged from 0 to 100, higher score is indicative of a higher response level (a high score for a symptom scale / item represents a high level of symptomatology / problems).
Time Frame: Baseline up to Cycle 60
Population: PRO evaluable population included participants from the safety analysis population who completed the assessments at baseline and at least one post-baseline time point. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Crizotinib 250 mg
Number analyzed (Participants) | 26
Units on a scale
  Dyspnea | -4.74 (14.791)
  Coughing | -12.82 (29.936)
  Hemoptysis | -5.12 (12.253)
  Sore mouth | -1.28 (14.844)
  Dysphagia | 0.00 (16.314)
  Peripheral neuropathy | 3.85 (19.611)
  Alopecia | -2.57 (20.910)
  Pain in chest | -12.82 (21.236)
  Pain in arm or shoulder | -15.37 (23.536)
  Pain in other parts | -7.68 (21.718)

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after the last dose of study treatment (maximum up to 295.9 weeks)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Crizotinib 250 mg
All-Cause Mortality (participants affected / at risk) | 65/127
Serious Adverse Events (participants affected / at risk) | 46/127
Other Adverse Events (participants affected / at risk) | 127/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crizotinib 250 mg (N=127)
Acute myocardial infarction (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Disease Progression (General disorders) | 7
Hepatic cyst (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2
Pneumonia (Infections and infestations) | 10
Appendicitis (Infections and infestations) | 1
Bronchiolitis (Infections and infestations) | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Empyema (Infections and infestations) | 1
Oesophageal infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Ruptured cerebral aneurysm (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Renal cyst (Renal and urinary disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Embolism (Vascular disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Bradycardia (Cardiac disorders) | 1
Retinal detachment (Eye disorders) | 1
Chronic gastritis (Gastrointestinal disorders) | 1
Hernia (General disorders) | 1
Peripheral swelling (General disorders) | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1
Liver injury (Hepatobiliary disorders) | 1
Postoperative wound infection (Infections and infestations) | 1
Renal tuberculosis (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Mediastinum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dysarthria (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Crizotinib 250 mg (N=127)
Neutropenia (Blood and lymphatic system disorders) | 14
Anaemia (Blood and lymphatic system disorders) | 15
Leukopenia (Blood and lymphatic system disorders) | 8
Sinus bradycardia (Cardiac disorders) | 11
Vision blurred (Eye disorders) | 25
Visual impairment (Eye disorders) | 22
Diplopia (Eye disorders) | 7
Photopsia (Eye disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 62
Nausea (Gastrointestinal disorders) | 58
Vomiting (Gastrointestinal disorders) | 50
Constipation (Gastrointestinal disorders) | 49
Abdominal pain upper (Gastrointestinal disorders) | 12
Abdominal pain (Gastrointestinal disorders) | 12
Stomatitis (Gastrointestinal disorders) | 10
Oedema peripheral (General disorders) | 39
Fatigue (General disorders) | 22
Pyrexia (General disorders) | 23
Chest pain (General disorders) | 11
Nasopharyngitis (Infections and infestations) | 28
Upper respiratory tract infection (Infections and infestations) | 22
Pneumonia (Infections and infestations) | 11
Urinary tract infection (Infections and infestations) | 11
Alanine aminotransferase increased (Investigations) | 72
Aspartate aminotransferase increased (Investigations) | 67
Neutrophil count decreased (Investigations) | 37
White blood cell count decreased (Investigations) | 30
Blood creatinine increased (Investigations) | 29
Gamma-glutamyltransferase increased (Investigations) | 18
Blood alkaline phosphate increased (Investigations) | 14
Decreased appetite (Metabolism and nutrition disorders) | 27
Hypoproteinaemia (Metabolism and nutrition disorders) | 14
Hypoalbuminaemia (Metabolism and nutrition disorders) | 18
Back pain (Musculoskeletal and connective tissue disorders) | 21
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16
Dysgeusia (Nervous system disorders) | 17
Dizziness (Nervous system disorders) | 23
Headache (Nervous system disorders) | 20
Insomnia (Psychiatric disorders) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 35
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12
Rash (Skin and subcutaneous tissue disorders) | 17
Pruritis (Skin and subcutaneous tissue disorders) | 11
Abdominal distension (Gastrointestinal disorders) | 8
Toothache (Gastrointestinal disorders) | 10
Asthenia (General disorders) | 9
Pain (General disorders) | 9
Peripheral swelling (General disorders) | 9
Hepatic function abnormal (Hepatobiliary disorders) | 10
Blood albumin decreased (Investigations) | 17
Blood creatine phosphokinase increased (Investigations) | 9
Protein total decreased (Investigations) | 7
Weight decreased (Investigations) | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 10
Hypokalaemia (Metabolism and nutrition disorders) | 10
Hyponatraemia (Metabolism and nutrition disorders) | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 10
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10
Hypoaesthesia (Nervous system disorders) | 7
Taste disorder (Nervous system disorders) | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 7

LIMITATIONS AND CAVEATS:
Due to small percentage of participants (less than 20%) after Cycle 60, data for EORTC QLQ-C30 score and EORTC QLQ-LC13 score could not be interpreted.

65 participants died during the whole study: 15 participants died within 28 days from last dose of study treatment and were reported as SAEs, while 50 participants died during the survival follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.